CLINICAL TRIAL: NCT06065423
Title: Evaluation of Home Program and Telerehabilitation for the Treatment Process in Patients With Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09.2021.131
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer Related Lymphedema; Telerehabilitation
MeSH Terms: conditions — Breast Cancer Lymphedema | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (Experimental): patients received exercises and massages through TR three times a week, conducted by a physiotherapist and a clinician. They were encouraged to perform their exercises and wear compression garments on the remaining days. Prior to the program, patients or their relatives received training from physiotherapists regarding exercises and Manual Lymphatic Drainage (MLD). Patients or their relatives were informed about the Zoom program and were instructed to acquire the application online. Two physiotherapists and groups of five patients each were organized based on rehabilitation days and hours, and access to the Zoom link was provided.
  Interventions: Other: Manuel Lymphatic Drainage(MLD), Exercises
- Home- Exercise Group (Active Comparator): patients were provided with a brochure explaining the massages and exercises they needed to perform. Additionally, they were contacted three times a week by a physiotherapist and a clinician to remind them of the treatments, assess the continuity and accuracy of the treatments, encourage them to perform the treatments correctly and consistently, and promote the wearing of compression garments.
  Interventions: Other: Manuel Lymphatic Drainage(MLD), Exercises

INTERVENTIONS:
Other: Manuel Lymphatic Drainage(MLD), Exercises — MLD:It is a unique massage technique that uses specific hand movements to provide a gentle pumping effect on the skin.
  Massage movements follow the direction of lymph flow and produce rapid results. The aim of this method is to achieve maximum skin tightening effect with minimum pressure.
  Exercise, on the other hand, increases physical performance, improves body composition, and provides an increase in quality of life by providing acute and chronic reductions in fatigue. Both aerobic exercises and strengthening exercises have been found effective on physical performance. It shows that a mixed program consisting of components such as aerobics, strengthening, coordination and stretching can positively affect flexibility, pain and energy expenditure in breast cancer patients.

SUMMARY:
During the Covid-19 pandemic, rehabilitation services for all patients were affected, and a term that was previously in use but gained popularity during the pandemic entered our vocabulary: 'Telerehabilitation'. The purpose of our study is to evaluate the treatment process and adherence of patients undergoing telerehabilitation.

DETAILED DESCRIPTION:
Our study is a randomized single-blind prospective study. Patients aged 18 to 75 years with stage 1-2 lymphedema associated with breast cancer and upper extremity lymphedema, who had undergone breast surgery at least 3 months prior, were included in the study. Group 1: Patients were given a brochure explaining the massage and exercises they should perform. They were periodically contacted by a physiotherapist and clinician to remind them of their tasks. Group 2: Patients underwent telerehabilitation exercises and massages three times a week guided by a physiotherapist and clinician, and on the remaining days, they continued their self-administered tasks. Patients were evaluated three times: before treatment, at weeks 5 and 8 after treatment. During each visit, patients' inter-limb volume difference, Quick DASH and Life Impact Scale scores, pain, tension, stiffness, and heaviness sensations were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone breast surgery at least 3 months ago
* Had stage 1-2 lymphedema
* Had upper extremity lymphedema associated with breast cancer

Exclusion Criteria:

* Signs of infection such as lymphangitis, cellulitis, fungal infections
* Those with documented lymph node metastases
* Those with bilateral lymphedema
* Those with other diseases affecting upper extremity functions
* Those with a history of previous surgery related to the upper extremity

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Volume Measurements | Time Frame: Day 0
  Arm measurement was measured with a tape measure at 4 cm intervals and calculated using the cone method in cm3
Volume Measurements | Time Frame: 5 weeks
  Arm measurement was measured with a tape measure at 4 cm intervals and calculated using the cone method in cm3
Volume Measurements | Time Frame: 8 weeks
  Arm measurement was measured with a tape measure at 4 cm intervals and calculated using the cone method in cm3
Symptom Severity | Time Frame: Day 0
  Shoulder pain, tightness, sensation of heaviness, and stiffness were evaluated using a numerical scale (1 to 10 points)
Symptom Severity | Time Frame: 5 weeks
  Shoulder pain, tightness, sensation of heaviness, and stiffness were evaluated using a numerical scale (1 to 10 points)
Symptom Severity | Time Frame: 8 weeks
  Shoulder pain, tightness, sensation of heaviness, and stiffness were evaluated using a numerical scale (1 to 10 points)
Functionality | Time Frame: Day 0
  Ouick Disabilities of the Arm, Shoulder and Hand (Quick DASH) questionnaire
Functionality | Time Frame: 5 weeks
  Ouick Disabilities of the Arm, Shoulder and Hand (Quick DASH) questionnaire
Functionality | Time Frame: 8 weeks
  Ouick Disabilities of the Arm, Shoulder and Hand (Quick DASH) questionnaire
Efficacity | Time Frame: Day 0
  Lymphedema Quality of Life Impact Scale
Efficacity | Time Frame: 5 weeks
  Lymphedema Quality of Life Impact Scale
Efficacity | Time Frame: 8 weeks
  Lymphedema Quality of Life Impact Scale

SECONDARY OUTCOMES:
Patient satisfaction with the treatment | Time Frame: 5 weeks
  Responses were gathered on a scale of very satisfied - satisfied - somewhat satisfied - unsatisfied
Patient satisfaction with the treatment | Time Frame: 8 weeks
  Responses were gathered on a scale of very satisfied - satisfied - somewhat satisfied - unsatisfied
patients were asked to compare their hand functionality to before the injury | Time Frame: 5 weeks
  Responses were gathered on a scale of 'much better - somewhat better - same - somewhat worse - much worse
patients were asked to compare their hand functionality to before the injury | Time Frame: 8 weeks
  Responses were gathered on a scale of 'much better - somewhat better - same - somewhat worse - much worse

CONTACTS AND LOCATIONS:
Overall Officials: CANAN ŞANAL TOPRAK, Study Director — Marmara University School of Medicine, Pendik Education and Research Hospital, Department of Physical Medicine and Rehabilitation
Locations (2):
- Turkey (Türkiye) (2):
  - Canan Şanal-Toprak, Istanbul
  - Marmara University School of Medicine, Pendik Education and Research Hospital, Department of Physical Medicine and Rehabilitation, Istanbul

IPD SHARING:
Plan to Share IPD: No